CLINICAL TRIAL: NCT00116584
Title: The Use of Heliox Driven Racemic Epinephrine Nebulization in the Treatment of Moderate to Severe Bronchiolitis in Pediatric Emergency Department Patients
Brief Title: Heliox-Driven Racemic Epinephrine in Treatment of Bronchiolitis in Pediatric ED Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Louisville (Other)
Responsible Party: Principal Investigator, In K. Kim, Professor, University of Louisville
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GRNT040954; GRNT040954; G040954 (Other Grant/Funding Number: Praxair Healthcare)
Record Dates: First submitted 2005-06-29; First posted 2005-06-30 (Estimated); Results first posted 2020-05-20 (Actual); Last update posted 2020-05-20 (Actual); Status verified 2020-05

CONDITIONS: Bronchiolitis
Keywords: heliox; bronchiolitis; racemic epinephrine
MeSH Terms: conditions — Bronchiolitis | interventions — heliox; Oxygen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- heliox (Other): heliox-driven nebulizations for children with moderate to severe bronchiolitis
  Interventions: Drug: heliox
- oxygen (Other): oxygen-driven nebulizations for children with moderate to severe bronchiolitis
  Interventions: Drug: oxygen

INTERVENTIONS:
Drug: heliox — continuous heliox therapy
  Arms: heliox
Drug: oxygen — continuous oxygen therapy
  Arms: oxygen

SUMMARY:
The purpose of this study is to assess whether children with moderate to severe bronchiolitis treated with standard racemic epinephrine therapy via 70:30 helium-oxygen (heliox) driven nebulization will have improvements in measurements of airway more rapidly than those treated with conventional air-oxygen driven nebulization.

ELIGIBILITY:
Inclusion Criteria:

* Any child 2-12 months old seen in the emergency department.
* A clinical bronchiolitis score > 3 by modified Wood's Clinical Bronchiolitis Score (M-WCBS).
* Diagnostic criteria of bronchiolitis includes tachypnea, cough, prolonged expiratory phase, wheezing, rales, chest retractions, and hyperinflation of lungs on chest radiograph. After consenting a patient to the study, respiratory syncytial virus (RSV) infection will be tested by rapid enzyme-linked immunoabsorbent assay of nasal secretions.

Exclusion Criteria:

* No child will be excluded based on race or gender
* Patients under the age of 2 months or greater than 12 months
* Patients with cyanotic heart disease
* Patients with lobar pneumonia, defined by results of chest radiographs.
* The presence of interstitial disease or diffuse patchy marking consistent with atelectasis on chest radiographs will not exclude patients.
* Patients with croup.
* Patients with foreign body aspiration.
* Patients with history of cystic fibrosis, bronchopulmonary dysplasia or other chronic lung disease.
* Patients with liver or renal disease.
* Patients with sickle cell anemia.
* Patients requiring mechanical ventilation.
* Patients who develop supraventricular tachycardia secondary to racemic epinephrine administration.
* Patients with tracheomalacia or bronchomalacia.
* Patients who had received bronchodilators within 2 hours of initiation of the study.
* Patients who had received systemic corticosteroids within 72 hours of enrollment
* Patients who suffered from persistent airway hyperreactivity in the 3 months before the study.
* Patients who do not tolerate the nasal cannulae for 45 out of 60 minutes.

Ages: 2 Months to 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 72 (Actual)
Dates: Start 2004-12; Primary Completion 2008-03 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: In K Kim, MD, Principal Investigator — University of Louisville, Dept. of Pediatrics, Div. of Pediatric Emergency Medicine
Locations (1):
- Kosair Children's Hospital, Louisville, Kentucky, United States

REFERENCES:
- [Result] Kim IK, Phrampus E, Sikes K, Pendleton J, Saville A, Corcoran T, Gracely E, Venkataraman S. Helium-oxygen therapy for infants with bronchiolitis: a randomized controlled trial. Arch Pediatr Adolesc Med. 2011 Dec;165(12):1115-22. doi: 10.1001/archpediatrics.2011.605. PMID 22147778

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted from October 1, 2004 through May 31, 2008 in the emergency department of an urban, tertiary care children's hospital.
Groups:
- Heliox: Patients were randomized to the helium-oxygen received nebulized racemic epinephrine via a face mask.
- Oxygen: Patients were randomized to 100% oxygen group and received nebulized racemic epinephrine via a face mask.
Period: Overall Study
Arm/Group | Heliox | Oxygen
Started | 36 | 36
Completed | 34 | 35
Not Completed | 2 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Protocol Violation | 1 | 1

BASELINE CHARACTERISTICS:
Population: Seventy-two subjects initially met inclusion criteria; but only 69 were in final analysis.
Groups:
- Oxygen: Oxygen nebulizations for children with moderate to severe bronchiolitis
- Total: Total of all reporting groups
Arm/Group | Heliox | Oxygen | Total
Number analyzed (Participants) | 34 | 35 | 69
Age, Continuous [Mean (Full Range); unit: Months] | 5.09 [2 to 12] | 6.11 [2 to 12] | 5.6 [2 to 12]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 11 | 22
  Male | 23 | 24 | 47

OUTCOME MEASURES:

1. Primary Outcome: Change in Modified Wood's Clinical Asthma Score (M-WCAS) From Baseline to 240 Minutes
Description: The Modified Wood's clinical Asthma Score is a score to measure severity of Asthma in children. There are 5 variables measured: oxygen saturation, inspiratory breath sounds, expiratory wheezing, accessory muscle involvement and cerebral function. Each variable is given a score of 0, 0.5, 1 or 2 with 2 being the most severe. The scores are combined from each variable to give a total. Total score ranges from 0 to 10, with a score of 10 (higher the score) indicating a worse outcome. We are reporting the degree of improvement in M-WCAS after assigned treatment.
Time Frame: 240 Minutes
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Heliox | Oxygen
Number analyzed (Participants) | 34 | 35
units on a scale | 1.84 [0 to 10] | .031 [0 to 10]
Statistical Analysis 1: Comparison: Heliox vs Oxygen; Test type: Superiority; p < 0.05, Fisher Exact

2. Secondary Outcome: Change in Modified Wood's Clinical Bronchiolitis Score (MWCBS) Between Oxygen and Heliox Groups at Various Times
Description: The Modified Wood's Clinical Bronchiolitis Score is based on a rating of saturated oxygen, inspiratory breath sounds, expiratory wheezing, accessory muscle use, cerebral function and wheezing. Each variable is rated 0, 0.5, 1, or 2. The total range of score is 0 to 2, with 2 (higher the score) indicating a worse outcome. For this outcome, a negative difference between groups represents an improvement.
Time Frame: 0, 60, 120, 180 and 240 min
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Heliox | Oxygen
Number analyzed (Participants) | 34 | 35
units on a scale
  Differenceof MWCBS at 0 mins | -0.33 [-0.71 to 0.59] | 0 [0 to 0]
  Difference of MWCBS at 60 mins | 0.54 [0.18 to 0.91] | 0 [0 to 0]
  Difference of MWCBS at 120 mins | 0.77 [0.45 to 1.09] | 0 [0 to 0]
  Difference of MWCBS at 180 mins | 0.94 [0.63 to 1.26] | 0 [0 to 0]
  Difference of MWCBS at 240 mins | 1.20 [0.87 to 1.54] | 0 [0 to 0]
Statistical Analysis 1: Comparison: Heliox vs Oxygen; Test type: Superiority; p < 0.05, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Change in Respiratory Distress Assessment Instrument (RDAI) Scores in Oxygen and Heliox Groups at Different Times
Description: The RDAI is an assessment instrument for respiratory distress. Patients are assigned a point value based on Wheezing (on expiration, inspiration and location) and Retractions (local of supraclavicular, intercostal and subcostal). Each subcategory is assigned a value of 0-4. The subscores are summed to give a total score for each variable (wheezing and retractions). The total score range for wheezing is 0 to 8, with 8 (higher the score) indicating a worse outcome. The total score range for retractions is 0 to 9, with 9 (higher the score) indicating a worse outcome. We are reporting the difference in score between the groups at various times, not a change from an earlier time. A positive value represents an improvement in the Heliox vs the Oxygen groups.
Time Frame: 0, 60, 120, 180 and 240 mins
Population: The Respiratory Distress Assessment Instrument (RDAI) has been used extensively. It is one of the most commonly used clinical scores for bronchiolitis,.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Heliox | Oxygen
Number analyzed (Participants) | 34 | 35
units on a scale
  Difference between RDAI at 0 min | -0.48 [-1.55 to 0.59] | 0 [0 to 0]
  Difference of RDAI at 60 mins | 1.80 [0.55 to 3.07] | 0 [0 to 0]
  Difference of RDAI at 120 mins | 2.92 [1.77 to 4.07] | 0 [0 to 0]
  Difference of RDAI at 180 mins | 3.00 [1.99 to 4.01] | 0 [0 to 0]
  Difference of RDAI at 240 mins | 3.29 [2.35 to 4.23] | 0 [0 to 0]
Statistical Analysis 1: Comparison: Heliox vs Oxygen; Test type: Superiority; p < 0.05, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Arm/Group | Heliox | Oxygen
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/35
Other Adverse Events (participants affected / at risk) | 0/34 | 0/35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No